CLINICAL TRIAL: NCT06427577
Title: Study on the Mechanism of ZhenQiFuZheng in the Treatment of Allergic Rhinitis Based on Intestinal Flora and Metabolites
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-304 ZhenQiFuZheng
Record Dates: First submitted 2024-04-26; First posted 2024-05-24 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allergic rhinitis (Experimental): ZhenQi FuZheng granules (ShiDaiYangGuang)
  1 bag at a time, twice a day. Oral for 4 weeks.
  Interventions: Drug: ZhenQi FuZheng granules (ShiDaiYangGuang)

INTERVENTIONS:
Drug: ZhenQi FuZheng granules (ShiDaiYangGuang) — 1 bag at a time, twice a day. Oral orally for 4 weeks.

SUMMARY:
ZhenQi FuZheng granules has been used to improve the immune function of human body, protect the bone marrow and adrenal cortex function and promote the recovery of positive function in traditional Chinese medicine care, especially with the immune imbalance diseases like post-surgery, chemotherapy and rhinitis. This project intends to establish AR（allergic rhinitis）specimen library, cell and animal model experiment, combining clinical cohort research with applied basic research, further assess the therapeutic mechanism of ZhenQiFuZheng granules in AR. We assume that ZhenQi FuZheng granules could cause the metabolic omics changes of nasal inflammatory factors and nasal secretions in AR patients, thus improving the type 2 inflammation level of allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-65 years).
* Patients who visited the Department of Otolaryngology of the First Affiliated Hospital of Nanjing Medical University and are diagnosed as allergic rhinitis .

Exclusion Criteria:

* Patients who refused to accept specimen and questionnaire collection.
* Patients who had nasal diseases other than allergic rhinitis, such as nasal papilloma and nasal malignant tumor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Rhinoconjunctivitis Quality of Life Questionnaire | 12 weeks
  Patients were scored by questionnaire before and after treatment, and the change in score before and after treatment was the primary outcome measure
Visual Analog Score for pain | 12 weeks
  Patients were scored by questionnaire before and after treatment, and the change in score before and after treatment was the primary outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Digheari A, Mahboub B, Tarraf H, Yucel T, Annesi-Maesano I, Doble A, Lahlou A, Tariq L, Aziz F, El Hasnaoui A. The clinical burden of allergic rhinitis in five Middle Eastern countries: results of the SNAPSHOT program. Allergy Asthma Clin Immunol. 2018 Nov 19;14:63. doi: 10.1186/s13223-018-0298-x. eCollection 2018. PMID 30473712
- [Background] Eifan AO, Durham SR. Pathogenesis of rhinitis. Clin Exp Allergy. 2016 Sep;46(9):1139-51. doi: 10.1111/cea.12780. PMID 27434218
- [Background] Cheng L, Chen J, Fu Q, He S, Li H, Liu Z, Tan G, Tao Z, Wang D, Wen W, Xu R, Xu Y, Yang Q, Zhang C, Zhang G, Zhang R, Zhang Y, Zhou B, Zhu D, Chen L, Cui X, Deng Y, Guo Z, Huang Z, Huang Z, Li H, Li J, Li W, Li Y, Xi L, Lou H, Lu M, Ouyang Y, Shi W, Tao X, Tian H, Wang C, Wang M, Wang N, Wang X, Xie H, Yu S, Zhao R, Zheng M, Zhou H, Zhu L, Zhang L. Chinese Society of Allergy Guidelines for Diagnosis and Treatment of Allergic Rhinitis. Allergy Asthma Immunol Res. 2018 Jul;10(4):300-353. doi: 10.4168/aair.2018.10.4.300. PMID 29949830
- [Background] Wang XD, Zheng M, Lou HF, Wang CS, Zhang Y, Bo MY, Ge SQ, Zhang N, Zhang L, Bachert C. An increased prevalence of self-reported allergic rhinitis in major Chinese cities from 2005 to 2011. Allergy. 2016 Aug;71(8):1170-80. doi: 10.1111/all.12874. Epub 2016 Apr 13. PMID 26948849
- [Background] Li K, Chen Y, Jiang R, Chen D, Wang H, Xiong W, Li D, Liu Z, Li X, Li J, Yuan K. Protective effects of astragaloside IV against ovalbumin-induced allergic rhinitis are mediated by T-box protein expressed in T cells/GATA-3 and forkhead box protein 3/retinoic acid-related orphan nuclear receptor gammat. Mol Med Rep. 2017 Aug;16(2):1207-1215. doi: 10.3892/mmr.2017.6685. Epub 2017 Jun 6. PMID 28586019